CLINICAL TRIAL: NCT06647108
Title: Randomized, Double-blind, Placebo-controlled Clinical Study to Evaluate the Effect of a Food Supplement on Apolipoprotein B in Individuals with Metabolic Syndrome Adhering to the Mediterranean Diet
Brief Title: Food Supplement for Individuals with Metabolic Syndrome
Acronym: META-TREAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ESI (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MetaTreat_RCT2024
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Apolipoprotein B; Dietary Supplement; Food Supplement; Mediterranean Diet; Body Composition
MeSH Terms: conditions — Metabolic Syndrome | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Food Supplement (Active Comparator): The composition of the dietary supplement is the following (for 1 sachet): 450 mg glucomannan, 250 mg white mulberry dry extract (d.e.), 200 mg gymnema (d.e.), 200 mg olive (d.e.), 200 mg Cassia nomame (d.e.), 200 mg Nopal, 5 mg policosanols and 20 µg chromium.
  Interventions: Dietary Supplement: Food Supplement
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Food Supplement — The composition of the dietary supplement is the following (for 1 sachet): 450 mg glucomannan, 250 mg white mulberry dry extract (d.e.), 200 mg gymnema (d.e.), 200 mg olive (d.e.), 200 mg Cassia nomame (d.e.), 200 mg Nopal, 5 mg policosanols and 20 µg chromium
  Arms: Food Supplement
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
In metabolic syndrome, blood levels of apolipoprotein B (Apo B) reveal the presence of quantitative and qualitative alterations of atherogenic lipoproteins and therefore represent an indicator of the risk of developing cardiovascular disease (CVD). The objective of this study is to evaluate the effect of a combined dietary supplement containing glucomannan, white mulberry dry extract (d.e.), gymnema (d.e.), olive (d.e.), Cassia nomame (d.e.), Nopal, policosanols and chromium, compared to placebo, on Apo B in individuals with metabolic syndrome adhering to the Mediterranean diet. Furthermore, the effect of the dietary supplement on anthropometric parameters, waist circumference and body composition will be investigated.

DETAILED DESCRIPTION:
Metabolic syndrome is a highly prevalent condition characterized by the simultaneous presence of multiple cardiometabolic risk factors, such as arterial hypertension, atherogenic dyslipidemia, hyperglycemia and abdominal obesity. According to the International Atherosclerosis Society (IAS), metabolic syndrome is a clustering of at least three of the following five medical conditions:

1. increased waist circumference (WC) (as per population- and country-specific definition)
2. increased levels of triglycerides (TG) (≥ 150 mg/dL)
3. reduced high-density lipoprotein cholesterol (HDL-C) levels (< 40 mg/dL in men and < 50 mg/dL in women)
4. increased blood pressure (BP) (systolic BP≥ 130 mmHg and/or diastolic BP≥ 85 mmHg)
5. impaired fasting glucose [fasting plasma glucose (FPG)≥ 100 mg/dL] In metabolic syndrome, blood levels of apolipoprotein B (Apo B) reveal the presence of quantitative and qualitative alterations of atherogenic lipoproteins and therefore represent an indicator of the risk of developing cardiovascular disease (CVD).

Troubling increases in high FPG, high body mass index (BMI), and other risk factors related to obesity and metabolic syndrome indicate an urgent need to identify and implement interventions, as shown by the Global Burden of Disease (GBD) Study Group. To date, several active ingredients of natural origin have been shown to favorably modify the individual components that have revealed the presence of metabolic syndrome. Among these, we find glucomannan and white mulberry dry extract.

The purpose of this study is to evaluate if a dietary supplement containing glucomannan, white mulberry dry extract (d.e.), gymnema (d.e.), olive (d.e.), Cassia nomame (d.e.), Nopal, policosanols and chromium, is able to significantly influence serum levels of apo B in individuals with metabolic syndrome adhering to the Mediterranean diet. Furthermore, the effect of the dietary supplement on anthropometric parameters, waist circumference and body composition will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years and ≤ 70 years old;
* Subjects with metabolic syndrome (according to the IAS criteria);
* Subjects with an estimated 10-year risk of CVD< 10% (as per the SCORE risk prediction algorithm of the ESC)
* Subjects who have the capability to communicate, to make themselves understood, and to comply with the study's requirements;
* Subjects agree to participate in the study and having dated and signed the informed consent form

Exclusion Criteria:

* Treatment with lipid-lowering drugs or taking food supplements that are effective on blood lipid levels;
* Chronic pharmacological treatments for any clinical condition not stabilized for at least 3 months;
* Known alterations in thyroid, renal or hepatic function (including transaminase values ≥ 3 times the times the upper limit of the normal range (ULN));
* Present or previous alcohol abuse;
* Pregnancy and breastfeeding;
* Subjects with known intolerance to one of the components of the tested dietary supplement;
* History or clinical evidence of any significant concomitant disease that could compromise the safety of the subject or the possibility of completing the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Effect of the Dietary Supplement on Apo B | From enrollment to the end of treatment at 12 weeks
  The primary objective is to compare the effect on Apo B after 12 weeks of treatment with the dietary supplement or placebo, in combination with the Mediterranean diet (Standard of Care - SOC).

SECONDARY OUTCOMES:
Effect of the Dietary Supplement on changes in body water | From enrollment to the end of treatment at 12 weeks
  To evaluate the effect of the dietary supplement on changes in body water compared baseline and placebo after 12 weeks of treatment.
Effect of the Dietary Supplement on changes in lean body mass | From enrollment to the end of treatment at 12 weeks
  To evaluate the effect of the dietary supplement on changes in lean body mass compared baseline and placebo after 12 weeks of treatment.
Effect of the Dietary Supplement on changes in fat body mass | From enrollment to the end of treatment at 12 weeks
  To evaluate the effect of the dietary supplement on changes in fat body mass compared baseline and placebo after 12 weeks of treatment.
Effect of the Dietary Supplement on changes in waist circumference | From enrollment to the end of treatment at 12 weeks
  To evaluate the effect of the dietary supplement on changes in waist circumference compared baseline and placebo after 12 weeks of treatment.
Dietary Supplement use and prevalence of Metabolic Syndrome | From enrollment to the end of treatment at 12 weeks
  To verify whether the intake of the dietary supplement is associated with a reduction in the prevalence of metabolic syndrome, compared to baseline and compared to placebo, after 12 weeks of treatment.
Effect of the Dietary Supplement on changes in body water midway through the study | From enrollment to 6-week follow-up
  To evaluate the effect of the dietary supplement on changes in body water compared baseline and placebo after 6 weeks of treatment
Effect of the Dietary Supplement on changes in lean body mass midway through the study | From enrollment to 6-week follow-up
  To evaluate the effect of the dietary supplement on changes in lean body mass compared baseline and placebo after 6 weeks of treatment.
Effect of the Dietary Supplement on changes in fat body mass effect on cholesterol midway through the study | From enrollment to 6-week follow-up
  To evaluate the effect of the dietary supplement on changes in fat body mass compared baseline and placebo after 6 weeks of treatment.
Effect of the Dietary Supplement on changes in waist circumference effect on cholesterol midway through the study | From enrollment to 6-week follow-up
  To evaluate the effect of the dietary supplement on changes in waist circumference compared baseline and placebo after 6 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Arrigo Francesco Giuseppe Cicero, MD, PhD, Principal Investigator — University of Bologna
Locations (1):
- IRCCS AOU di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No